CLINICAL TRIAL: NCT06770621
Title: Longitudinal Study of the GLUcagon REsponse to Hypoglycemia in Children and Adolescents With New-onset Type 1 DIAbetes (GLUREDIA Study): Characteristics and Predictive Biomarkers.
Brief Title: Longitudinal Study of the GLUcagon REsponse to Hypoglycemia in Children and Adolescents With New-onset Type 1 DIAbetes
Acronym: GLUREDIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/02FEV/043
Record Dates: First submitted 2024-07-25; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Severe Hypoglycemia; Type1diabetes
Keywords: Pediatric; Hypoglycemia; Diabetes
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Interventional study, parallel Assignment, the main objective is diagnostic, open-label, this study has 7 sub-sections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- To investigate the evolution of pancreatic α-cell function. (WP1) (Experimental): Regular clinical and biological monitoring will be conducted during this period, as well as four insulin-induced hypoglycemia (IIH) tests. Hormones and other blood parameters will be measured, and an analysis of the genome, proteome, and micro-RNAs (miRs) will be performed during these IIH tests and throughout the biological monitoring. The primary goal of this study is to find a correlation between the patient's phenotype and the various biological results obtained, mainly blood biomarkers, in order to subsequently determine models to predict the state of pancreatic α-cell function in the first months post-diagnosis.
  Interventions: Diagnostic Test: Insulin-induced hypoglycemia test
- Conduct an assessment of the management of severe hypoglycemia. (WP2) (Active Comparator): Study of glycemic variations collected by the continuous glucose monitoring sensor in the days preceding a severe hypoglycemia. The aim of this analysis is to identify a specific glycemic profile in patients in the days leading up to severe hypoglycemia in order to better anticipate such events.
  Interventions: Other: Observation-questionnaire
- Evaluate the α-cell function in first-degree relatives of patients with type 1 diabetes. (WP3) (Experimental): In this cohort of relatives, the investigators will evaluate the function of pancreatic α-islets and the counter-regulation mechanism. This evaluation will have two main objectives. The first objective will be to compare this counter-regulation mechanism between individuals without type 1 diabetes and patients with type 1 diabetes. The second objective is to determine whether the dysfunction of the counter-regulation mechanism in diabetic patients is solely due to type 1 diabetes or if there is a familial component to this dysfunction.
  Interventions: Diagnostic Test: Insulin-induced hypoglycemia test
- Characterize the glycemic profile and α-cell function. (WP4) (Experimental): The aim is to assess residual function in patients with pancreatic disease, the phenomenon of counter-regulation and its impact on carbohydrate metabolism. To this end, IIH tests will be carried out in these patients, during which blood samples will be taken as in patients with type 1 diabetes (see above). This group of patients will also serve as a control group for the study of our diabetic patients.
  Patient with : exocrine dysfunction of the pancreas either as a consequence of cystic fibrosis or as a consequence of (sub)total pancreatectomy.
  Interventions: Diagnostic Test: Insulin-induced hypoglycemia test
- Evaluate the phenomenon of counter-regulation in patients with proven growth hormone. (WP5) (Active Comparator): These patients will serve as control groups for our GLUREDIA study to assess counter-regulation in our diabetic patients.
  Patient with : groth hormone or adrenal hormone deficiency and in healthy patients with no proven hormone deficiency.
  Interventions: Diagnostic Test: Insulin-induced hypoglycemia test
- Study the link between the clinical characteristics of diabetic patients and their genome (WP6) (Experimental): For each participant, the investigators will study their clinical history and the evolution of their glycemic parameters from diagnosis to the date they agreed to take part in the study (retrospective analysis). Next, each patient's exome will be analyzed from a blood tube taken during a consultation following agreement to take part in the study. With these analyses, the investigators hope to gain a better understanding of the clinical course of our diabetic patients and their risk of severe hypoglycemia.
  Interventions: Other: Biological sample once
- Evaluation of the circadian rhythm of glucagon (WP7) (Experimental): After recruitment, each participant will complete a questionnaire assessing their sensitivity to hypoglycemia. Based on their responses and phenotype, participants will be divided into two cohorts for analysis. Subsequently, a glucagon profile will be established for each participant through quarterly consultations involving blood samples taken by a pediatric nurse.
  Interventions: Diagnostic Test: Glucagon profile

INTERVENTIONS:
Diagnostic Test: Insulin-induced hypoglycemia test — For these tests, multiple blood samples will be collected during insulin-induced hypoglycemia (stage 1 hypoglycemia is defined as a blood glucose level below 70 mg/dL, while stage 2 corresponds to values below 54 mg/dL). The tests will be conducted on patients who have fasted for at least 12 hours and will be supervised by a medical staff member trained to manage severe hypoglycemia.
  Arms: Characterize the glycemic profile and α-cell function. (WP4); Evaluate the phenomenon of counter-regulation in patients with proven growth hormone. (WP5); Evaluate the α-cell function in first-degree relatives of patients with type 1 diabetes. (WP3); To investigate the evolution of pancreatic α-cell function. (WP1)
Diagnostic Test: Glucagon profile — The subject must fast before the consultation and follow a specific diet the day before; after an initial blood draw (P1), the patient will have breakfast and take any required insulin, followed by two additional blood draws 1.5 hours after breakfast (P2) and 1.5 hours after P2 (P3)
  Arms: Evaluation of the circadian rhythm of glucagon (WP7)
Other: Biological sample once — The exome of each patient will then be analyzed from the blood sample taken beforehand.
  Arms: Study the link between the clinical characteristics of diabetic patients and their genome (WP6)
Other: Observation-questionnaire — only the answer to a questionnaire
  Arms: Conduct an assessment of the management of severe hypoglycemia. (WP2)

SUMMARY:
The GLUREDIA study investigates the counter-regulatory response (CRR) during hypoglycemia in children with type 1 diabetes (T1D). Hypoglycemia can lead to severe symptoms, but is normally counteracted by CRR, corresponding to the secretion of hormones to maintain normoglycemia. Hypoglycemia is common in T1DM but some patients develop severe hypoglycemia as a result of CRR dysfunction. Despite several studies in adults, the presence of CRR dysfunction remains unpredictable and not well understood. The objective of GLUREDIA is therefore to describe and predict the evolution of CRR in children with T1DM.

ELIGIBILITY:
WP1 :

* Inclusion criteria:

  * De novo type 1 diabetic patient, as per ISPAD criteria;
  * Symptoms of hyperglycemia: polyuria-polydipsia-amaigrin +/- Acido ketosis.
  * Fasting blood glucose ≥126 mg/dL AND/OR blood glucose ≥200 mg/dL at 120 minutes of an OGTT AND/OR HbA1c ≥6.5% AND/OR a patient with symptoms of hyperglycemia/hyperglycemic crisis (see 8. a. 2.) with random blood glucose ≥200 mg/dL.

Presence in serum of one or more anti-islet autoantibodies (anti-insulin, anti-IA2, anti-GAD65, anti-ZnT8)

* Patients aged between 2 and 30 years
* Minimum weight: 17 kg (for blood samples)
* Male - female patients
* Free, written and oral consent.

  * Exclusion criteria:
* Child under 2 years of age.
* Taking treatments interfering with insulin secretion and sensitivity (e.g. sulfonylureas, diazoxide, somatostatin, methylxanthine derivatives, corticosteroids, biguanide, incretins).
* Presence of newly diagnosed (within 1 month) celiac disease (diagnosed on pathological duodenal biopsy) at inclusion.
* Autoimmune/autoinflammatory disease (other than type 1 diabetes) or active malignancy present at inclusion.
* Obesity defined as a BMI with a z-score >+3 SD.
* Hepatic, renal or adrenal insufficiency.
* History of bone marrow transplantation.
* History of diabetes after hemolytic-uremic syndrome.
* Epileptic patient
* Absence of anti-islet autoantibodies.
* Dysmorphia with suspicion of underlying genetic syndrome.
* Participation in another study in the previous 3 months, with administration of blood derivatives or potentially immunomodulating treatments.

WP2 :

* Inclusion Criteria:

  * De novo type 1 diabetic patient, as per ISPAD criteria;
  * Symptoms of hyperglycemia: polyuria-polydipsia-amaigrin +/- Acido ketosis.
  * Fasting blood glucose ≥126 mg/dL AND/OR blood glucose ≥200 mg/dL at 120 minutes of an OGTT AND/OR HbA1c ≥6.5% AND/OR a patient with symptoms of hyperglycemia/hyperglycemic crisis (see 8. a. 2.) with random blood glucose ≥200 mg/dL.
  * Presence in serum of one or more anti-islet autoantibodies (anti-insulin, anti-IA2, anti-GAD65, anti-ZnT8)
  * Patients aged between 2 years and 18 years (<18 years).
  * Male - female patients
  * Free, written and oral consent.
* Exclusion criteria:

  * Child under 2 years of age.
  * Taking treatments that interfere with insulin secretion and sensitivity (e.g. sulfonylureas, diazoxide, somatostatin, methylxanthine derivatives, corticosteroids, biguanide, incretins).
  * Presence of newly diagnosed (within 1 month) celiac disease (diagnosed on pathological duodenal biopsy) at inclusion.
  * Autoimmune/autoinflammatory disease (other than type 1 diabetes) or active malignancy present at inclusion.
  * Obesity defined as a BMI with a z-score >+3 SD.
  * Hepatic, renal or adrenal insufficiency.
  * History of bone marrow transplantation.
  * History of diabetes after hemolytic-uremic syndrome.
  * Absence of anti-islet autoantibodies.
  * Dysmorphia with suspected underlying genetic syndrome.
  * Participation in another study within the previous 3 months with administration of blood derivatives or potentially immunomodulatory treatments.

WP3 :

* Inclusion Criteria:

  * Adult older than 18 years.
  * Absence of blood marker of diabetes (Absence of antibodies, HbA1C <6.5%, C-peptide > 0.18 nmol/L, Fasting blood glucose < 100 mg/dL, blood glucose at any time < 200 mg/dL).
  * Be a first-degree relative with a patient being followed for diabetes (meeting ISPAD criteria).
  * Male - Female
  * Free written and oral consent
* Exclusion criteria:

  * Taking treatments that interfere with insulin secretion and sensitivity (e.g. sulfonylureas, diazoxide, somatostatin, methylxanthine derivatives, corticosteroids, biguanide, incretins).
  * Presence of newly diagnosed (within 1 month) celiac disease (diagnosed on pathological duodenal biopsy) at inclusion.
  * Autoimmune/autoinflammatory disease (other than type 1 diabetes) or active malignancy present at inclusion.
  * Obesity defined as a BMI with a z-score >+3 SD.
  * Hepatic, renal or adrenal insufficiency.
  * History of bone marrow transplantation.
  * History of diabetes after hemolytic-uremic syndrome.
  * Ischemic cardiomyopathy
  * Pregnant participant
  * Epileptic patient

WP4 :

* Inclusion Criteria:

Cohort of patients followed for cystic fibrosis:

* Pediatric patient between 2 and 18 years of age.
* Diagnosed with cystic fibrosis with impaired pancreatic endocrine function.
* Presents glucose homeostasis disorders (regular hypo/hyper-glycemia).
* Male - female patient
* Free, written and oral consent

Cohort of patients with (sub)total pancreatectomy:

* Pediatric patients between 2 and 18 years of age.
* Follow-up for total pancreatectomy or caudal pancreatectomy
* Presents disorders of carbohydrate homeostasis (regular hypo-/hyper-glycemia)
* Male - female patient
* Free, written and oral consent

  * Exclusion criteria:
* Child under 2 years of age.
* Body weight less than 17 kg.
* Taking treatments that interfere with insulin secretion and sensitivity (e.g. sulfonylureas, diazoxide, somatostatin, methylxanthine derivatives, corticosteroids, biguanide, incretins).
* Presence of newly diagnosed (within 1 month) celiac disease (diagnosed on pathological duodenal biopsy) at inclusion.
* Autoimmune/autoinflammatory disease (other than type 1 diabetes) or active malignancy present at inclusion.
* Obesity defined as a BMI with a z-score >+3 SD.
* Hepatic, renal or adrenal insufficiency.
* History of bone marrow transplantation.
* History of diabetes after hemolytic-uremic syndrome.
* Dysmorphia with suspected underlying genetic syndrome.
* Participation in another study within the last 3 months, with administration of blood derivatives or potentially immunomodulatory treatments.

WP5 :

* Inclusion Criteria:

  * Patient who has undergone insulin testing due to suspected growth hormone deficiency or adrenal insufficiency or hypopituitarism.
  * Patients between the ages of 2 years and 18 years (<18 years).
  * Male - female patient.
  * Free written and oral consent.
* Exclusion criteria:

  * Child under 2 years of age.
  * Body weight less than 17 kg.
  * Taking treatments that interfere with insulin secretion and sensitivity (e.g. sulfonylureas, diazoxide, somatostatin, methylxanthine derivatives, corticosteroids, biguanide, incretins).
  * Presence of newly diagnosed (within 1 month) celiac disease (diagnosed on pathological duodenal biopsy) at inclusion.
  * Autoimmune/autoinflammatory disease (other than type 1 diabetes) or active malignancy present at inclusion.
  * Obesity defined as a BMI with a z-score >+3 SD..
  * History of bone marrow transplantation.
  * History of diabetes after hemolytic-uremic syndrome.
  * Participation in another study within the last 3 months, with administration of blood derivatives or potentially immunomodulatory treatments.

WP6 :

* Inclusion Criteria:

  * Type 1 diabetic patient, as per ISPAD criteria;
  * Symptoms of hyperglycemia: polyuria-polydipsia-amaigrin +/- Acido ketosis.
  * Fasting blood glucose ≥126 mg/dL AND/OR blood glucose ≥200 mg/dL at 120 minutes of an OGTT AND/OR HbA1c ≥6.5% AND/OR a patient with symptoms of hyperglycemia/hyperglycemic crisis (see 8. a. 2.) with random blood glucose ≥200 mg/dL.
  * Presence in serum of one or more anti-islet autoantibodies (anti-insulin, anti-IA2, anti-GAD65, anti-ZnT8)
  * Patients aged between 2 and 18 years (<18 years).
  * Male - female patients
  * Free, written and oral consent.
* Exclusion criteria:

  * Child under 2 years of age.
  * Taking treatments interfering with insulin secretion and sensitivity (e.g. sulfonylureas, diazoxide, somatostatin, methylxanthine derivatives, corticosteroids, biguanide, incretins).
  * Autoimmune/autoinflammatory disease (other than type 1 diabetes) or active malignancy present at inclusion.
  * Obesity defined as a BMI with a z-score >+3 SD.
  * Hepatic, renal or adrenal insufficiency.
  * History of bone marrow transplantation.
  * History of diabetes after hemolytic-uremic syndrome.
  * Epileptic patient
  * Dysmorphia with suspicion of underlying genetic syndrome.
  * Participation in another study in the previous 3 months, with administration of blood derivatives or potentially immunomodulating treatments.

WP7 :

* Inclusion Criteria:

  * De novo type 1 diabetic patient, as per ISPAD criteria;
  * Symptoms of hyperglycemia: polyuria-polydipsia-amaigrin +/- Acido ketosis.
  * Fasting blood glucose ≥126 mg/dL AND/OR blood glucose ≥200 mg/dL at 120 minutes of an OGTT AND/OR HbA1c ≥6.5% AND/OR a patient with symptoms of hyperglycemia/hyperglycemic crisis (see 8. a. 2.) with random blood glucose ≥200 mg/dL.
  * Presence in serum of one or more anti-islet autoantibodies (anti-insulin, anti-IA2, anti-GAD65, anti-ZnT8)
  * Patients aged between 2 and 18 years
  * Minimum weight: 17 kg (for blood samples)
  * Male - female patients
  * Free, written and oral consent.
* Exclusion criteria:

  * Child under 2 years of age.
  * Taking treatments interfering with insulin secretion and sensitivity (e.g. sulfonylureas, diazoxide, somatostatin, methylxanthine derivatives, corticosteroids, biguanide, incretins).
  * Presence of newly diagnosed (within 1 month) celiac disease (diagnosed on pathological duodenal biopsy) at inclusion.
  * Autoimmune/autoinflammatory disease (other than type 1 diabetes) or active malignancy present at inclusion.
  * Obesity defined as a BMI with a z-score >+3 SD.
  * Hepatic, renal or adrenal insufficiency.
  * History of bone marrow transplantation.
  * History of diabetes after hemolytic-uremic syndrome.
  * Epileptic patient
  * Absence of anti-islet autoantibodies.
  * Dysmorphia with suspicion of underlying genetic syndrome.
  * Participation in another study in the previous 3 months, with administration of blood derivatives or potentially immunomodulating treatments.

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
To investigate the evolution of pancreatic α-cell function. (WP1) | 18 months per patient
  Regular clinical and biological monitoring will be performed during this period as well as four insulin-induced hypoglycemia (IIH) tests.
To evaluate the presence of blood biomarkers that correlate with the evolution of α-cell function. (WP1) | 18 months per patient
  Regular clinical and biological monitoring will be performed during this period as well as four insulin-induced hypoglycemia (IIH) tests. Hormones and other blood parameters will be measured and genome, proteome and microRNA (miRs) analysis will be performed during the IIH tests and during the biological follow-up. The expected results are the description and prediction of CRR in the first months after T1DM.

SECONDARY OUTCOMES:
Conduct an assessment of the management of severe hypoglycemia. (WP2) | Baseline
  Use of a questionnaire which is sent out once per patient during a routine consultation. The analysis does not take the form of a score, but is based on the analysis of the answers to the question according to the patient's profile. (WP2)
Evaluate the α-cell function in first-degree relatives of patients with type 1 diabetes. (WP3) | Baseline
  In the remaining parents, those without biological signs of (pre-)diabetes, an IIH test will be performed during which blood samples identical to those performed in patients with type 1 diabetes will be taken. (WP3)
Characterize the glycemic profile and α-cell function. (WP4) | Baseline
  IIH tests will be performed in these patients during which blood samples will be taken as in patients with type 1 diabetes. This group of patients will also be a control group for the study of our diabetic patients. (WP4)
Evaluate the phenomenon of counter-regulation in patients with proven growth hormone. (WP5) | Baseline
  Patients suspected of adrenal or pituitary hormone deficiency, will perform as part of their diagnosis a hypoglycemic test. Here the difference is that the investigators will add two additional tubes to each sample, to those already collected as part of the hypoglycemic test. These tubes will be used, as in the other parts, to measure hormones and other blood parameters, as well as to perform an analysis of the genome, proteome and micro-RNAs (miRs).
  (WP5)
Study the link between the clinical characteristics of diabetic patients and their genome (WP6) | Baseline
  For each participant, the investigators will study their clinical history, the evolution of their glycemic parameters from diagnosis to the date they agree to take part in the study (retrospective analysis). Next, each patient's exome will be analyzed from a blood tube taken during a consultation following agreement to take part in the study. With these analyses, the inestigators hope to gain a better understanding of the clinical course of our diabetic patients and their risk of severe hypoglycemia. (WP6)
Evaluation of the circadian rhythm of glucagon (WP7) | Baseline
  Each participant will complete a questionnaire assessing his or her susceptibility to hypoglycemia. A glucagonemic profile will then be established for each participant. This step, carried out during quarterly consultations, will involve blood sampling. (WP7)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lysy, Pr, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Clinique Universitaires Saint Luc, Brussels, Woluwe-saint-lambert, Belgium

IPD SHARING:
Plan to Share IPD: No